CLINICAL TRIAL: NCT05886699
Title: Comparison of Efficacy of Autologous Platelet - Rich Plasma Combined With Demineralized Freeze - Dried Bone Allograft Versus Demineralized Freeze - Dried Bone Allograft: A Randomized Clinical Trial in Central India
Brief Title: Comparison of PRP & DFDBA vs. DFDBA in Intrabony Periodontal Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government Dental College and Hospital, India (Other Government)
Responsible Party: Principal Investigator, Dr. Pallavi Meshram, Assistant Professor, Government Dental College and Hospital, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PMeshram
Record Dates: First submitted 2015-03-02; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Chronic Periodontitis
Keywords: platelet - rich plasma; demineralized freeze - dried bone allograft; intrabony defect; periodontitis.
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRP combined with DFDBA (Experimental): Open flap debridement, followed by placement of PRP combined with DFDBA
  Interventions: Other: PRP combined with DFDBA
- DFDBA (Active Comparator): Open flap debridement, followed by placement of DFDBA
  Interventions: Other: DFDBA

INTERVENTIONS:
Other: PRP combined with DFDBA — Periodontal intrabony defects were treated with open flap debridement followed by placement of PRP combined with DFDBA
  Arms: PRP combined with DFDBA
Other: DFDBA — Periodontal intrabony defects were treated with open flap debridement followed by placement of PRP combined with DFDBA
  Arms: DFDBA

SUMMARY:
The purpose of this clinical trial is to compare the results in subjects with periodontitis using subjects own blood - Platelet-rich plasma (PRP) combined with bone graft material, namely, Demineralized Freeze - Dried Bone Allograft (DFDBA) or DFDBA alone in the treatment of bone defects around the teeth.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, 13 patients giving written informed consent and who meet the eligibility requirements were randomly allocated in a single blind manner (participants) to test group (PRP combined with DFDBA) or control group (DFDBA).

33 sites (18 test, 15 control unpaired defects) were treated - 1) to investigate the possible additional effects of PRP when combined with DFDBA, and 2) to compare the clinical and radiographic outcomes obtained in test and control groups,12 months post - operatively.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* with chronic periodontitis
* who were free of local or systemic disease
* who had not received any type of periodontal therapy in the last six months
* radiograph showing at least one angular defect in any quadrant
* the involved teeth were vital and asymptomatic
* the site of interest had at least 2 mm of keratinized gingiva on the facial aspect of the selected teeth

Exclusion Criteria:

* Patients with abnormal platelet count
* allergic to chlorhexidine or any other medicine used in the study
* showing unacceptable oral hygiene compliance during / after the phase I therapy;
* pregnant or lactating mothers;
* smokers
* endodontically involved teeth
* patients under any medication known to interfere with periodontal healing. e.g., corticosteroids
* on anticoagulant therapy
* patients with transferable jobs or who were uncooperative
* patients participating in other dental clinical trials.

Ages: 28 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in Probing Pocket Depth (PPD) from baseline to 12 months | baseline to 12 months
  PPD is vertical measurement from the free gingival margin to the base of the pocket measured to the nearest millimeter using a UNC (University of North Carolina) -15 periodontal probe.
Change in Periodontal Attachment Level (PAL) from baseline to 12 months | baseline to 12 months
  PAL is vertical measurement recorded with the help of customized acrylic stent from a fixed reference point to the base of the pocket measured to the nearest millimeter using UNC - 15 probe
Change in Gingival Recession (GR) from baseline to 12 months | baseline to 12 months
  GR is vertical measurement recorded with the help of customized acrylic stent from a fixed reference point to the gingival margin measured to the nearest millimeter using UNC-15 probe
Change in Crestal bone resorption from baseline to 12 months | baseline to 12 months
  Crestal bone resorption is the distance from Cementoenamel Junction to the Alveolar Crest (CEJ- AC); measured in millimeters using standardized intraoral periapical (IOPA) radiographs along with a calibrated grid of the tooth of interest
Change in Defect fill from baseline to 12 months | baseline to 12 months
  Defect fill is the distance from Cementoenamel Junction to Base of the Defect (CEJ- BD); measured in millimeters using standardized intraoral periapical (IOPA) radiographs along with a calibrated grid of the tooth of interest
Change in Defect resolution from baseline to 12 months | baseline to 12 months
  Defect resolution is the distance from the Alveolar Crest to Base of the Defect (AC - BD); measured in millimeters using standardized intraoral periapical (IOPA) radiographs along with a calibrated grid of the tooth of interest

SECONDARY OUTCOMES:
Plaque Index | baseline to 12 months
  Silness and Loe, 1964
Gingival Index | baseline to 12 months
  Loe and Silness, 1963

CONTACTS AND LOCATIONS:
Overall Officials: Pallavi A Meshram, MDS, Principal Investigator — Government Dental College and Hospital, Nagpur, India; Ramreddy K Yeltiwar, MDS, Study Chair — Rungta College of Dental Sciences and Research, Bhilai, India.; Mangesh B Phadnaik, MDS, Study Director — Government Dental College and Hospital, Nagpur, India
Locations (1):
- 212, Department of Periodontology, Government Dental college and Hospital, Nagpur, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Yes
All collected Individual Participant Data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: to other researchers

REFERENCES:
- [Background] Pihlstrom BL, Michalowicz BS, Johnson NW. Periodontal diseases. Lancet. 2005 Nov 19;366(9499):1809-20. doi: 10.1016/S0140-6736(05)67728-8. PMID 16298220
- [Background] Polimeni G, Xiropaidis AV, Wikesjo UM. Biology and principles of periodontal wound healing/regeneration. Periodontol 2000. 2006;41:30-47. doi: 10.1111/j.1600-0757.2006.00157.x. No abstract available. PMID 16686925
- [Background] Quintero G, Mellonig JT, Gambill VM, Pelleu GB Jr. A six-month clinical evaluation of decalcified freeze-dried bone allografts in periodontal osseous defects. J Periodontol. 1982 Dec;53(12):726-30. doi: 10.1902/jop.1982.53.12.726. PMID 6759628
- [Background] Rummelhart JM, Mellonig JT, Gray JL, Towle HJ. A comparison of freeze-dried bone allograft and demineralized freeze-dried bone allograft in human periodontal osseous defects. J Periodontol. 1989 Dec;60(12):655-63. doi: 10.1902/jop.1989.60.12.655. PMID 2693682
- [Background] Gajiwala AL, Kumar BD, Chokhani P. Evaluation of demineralised, freeze-dried, irradiated bone allografts in the treatment of osseous defects in the oral cavity. Cell Tissue Bank. 2007;8(1):23-30. doi: 10.1007/s10561-006-9014-z. PMID 16838195
- [Background] Mellonig JT. Autogenous and allogeneic bone grafts in periodontal therapy. Crit Rev Oral Biol Med. 1992;3(4):333-52. doi: 10.1177/10454411920030040201. PMID 1391415
- [Background] Marx RE, Carlson ER, Eichstaedt RM, Schimmele SR, Strauss JE, Georgeff KR. Platelet-rich plasma: Growth factor enhancement for bone grafts. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1998 Jun;85(6):638-46. doi: 10.1016/s1079-2104(98)90029-4. PMID 9638695
- [Background] Demir B, Sengun D, Berberoglu A. Clinical evaluation of platelet-rich plasma and bioactive glass in the treatment of intra-bony defects. J Clin Periodontol. 2007 Aug;34(8):709-15. doi: 10.1111/j.1600-051X.2007.01108.x. PMID 17635247
- [Background] Camargo PM, Lekovic V, Weinlaender M, Vasilic N, Madzarevic M, Kenney EB. Platelet-rich plasma and bovine porous bone mineral combined with guided tissue regeneration in the treatment of intrabony defects in humans. J Periodontal Res. 2002 Aug;37(4):300-6. doi: 10.1034/j.1600-0765.2002.01001.x. PMID 12200975
- [Background] Lekovic V, Camargo PM, Weinlaender M, Vasilic N, Kenney EB. Comparison of platelet-rich plasma, bovine porous bone mineral, and guided tissue regeneration versus platelet-rich plasma and bovine porous bone mineral in the treatment of intrabony defects: a reentry study. J Periodontol. 2002 Feb;73(2):198-205. doi: 10.1902/jop.2002.73.2.198. PMID 11895286
- [Background] de Obarrio JJ, Arauz-Dutari JI, Chamberlain TM, Croston A. The use of autologous growth factors in periodontal surgical therapy: platelet gel biotechnology--case reports. Int J Periodontics Restorative Dent. 2000 Oct;20(5):486-97. PMID 11203586
- [Background] Piemontese M, Aspriello SD, Rubini C, Ferrante L, Procaccini M. Treatment of periodontal intrabony defects with demineralized freeze-dried bone allograft in combination with platelet-rich plasma: a comparative clinical trial. J Periodontol. 2008 May;79(5):802-10. doi: 10.1902/jop.2008.070436. PMID 18454658
- [Background] Armitage GC. Development of a classification system for periodontal diseases and conditions. Ann Periodontol. 1999 Dec;4(1):1-6. doi: 10.1902/annals.1999.4.1.1. PMID 10863370
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Background] Pradeep AR, Shetty SK, Garg G, Pai S. Clinical effectiveness of autologous platelet-rich plasma and Peptide-enhanced bone graft in the treatment of intrabony defects. J Periodontol. 2009 Jan;80(1):62-71. doi: 10.1902/jop.2009.080214. PMID 19228091
- [Background] Hanna R, Trejo PM, Weltman RL. Treatment of intrabony defects with bovine-derived xenograft alone and in combination with platelet-rich plasma: a randomized clinical trial. J Periodontol. 2004 Dec;75(12):1668-77. doi: 10.1902/jop.2004.75.12.1668. PMID 15732870
- [Background] Gonshor A. Technique for producing platelet-rich plasma and platelet concentrate: background and process. Int J Periodontics Restorative Dent. 2002 Dec;22(6):547-57. PMID 12516826
- [Background] Sharma A, Pradeep AR. Treatment of 3-wall intrabony defects in patients with chronic periodontitis with autologous platelet-rich fibrin: a randomized controlled clinical trial. J Periodontol. 2011 Dec;82(12):1705-12. doi: 10.1902/jop.2011.110075. Epub 2011 Apr 5. PMID 21513477
- [Background] Linares A, Cortellini P, Lang NP, Suvan J, Tonetti MS; European Research Group on Periodontology (ErgoPerio). Guided tissue regeneration/deproteinized bovine bone mineral or papilla preservation flaps alone for treatment of intrabony defects. II: radiographic predictors and outcomes. J Clin Periodontol. 2006 May;33(5):351-8. doi: 10.1111/j.1600-051X.2006.00911.x. PMID 16634957
- [Background] Cortellini P, Prato GP, Tonetti MS. The simplified papilla preservation flap. A novel surgical approach for the management of soft tissues in regenerative procedures. Int J Periodontics Restorative Dent. 1999 Dec;19(6):589-99. PMID 10815597
- [Background] Camargo PM, Lekovic V, Weinlaender M, Vasilic N, Madzarevic M, Kenney EB. A reentry study on the use of bovine porous bone mineral, GTR, and platelet-rich plasma in the regenerative treatment of intrabony defects in humans. Int J Periodontics Restorative Dent. 2005 Feb;25(1):49-59. PMID 15736778
- [Background] Okuda K, Tai H, Tanabe K, Suzuki H, Sato T, Kawase T, Saito Y, Wolff LF, Yoshiex H. Platelet-rich plasma combined with a porous hydroxyapatite graft for the treatment of intrabony periodontal defects in humans: a comparative controlled clinical study. J Periodontol. 2005 Jun;76(6):890-8. doi: 10.1902/jop.2005.76.6.890. PMID 15948682
- [Background] Christgau M, Moder D, Wagner J, Glassl M, Hiller KA, Wenzel A, Schmalz G. Influence of autologous platelet concentrate on healing in intra-bony defects following guided tissue regeneration therapy: a randomized prospective clinical split-mouth study. J Clin Periodontol. 2006 Dec;33(12):908-21. doi: 10.1111/j.1600-051X.2006.00999.x. PMID 17092242
- [Background] Dori F, Huszar T, Nikolidakis D, Arweiler NB, Gera I, Sculean A. Effect of platelet-rich plasma on the healing of intra-bony defects treated with a natural bone mineral and a collagen membrane. J Clin Periodontol. 2007 Mar;34(3):254-61. doi: 10.1111/j.1600-051X.2006.01044.x. Epub 2007 Jan 25. PMID 17257158
- [Background] Okuda K, Kawase T, Momose M, Murata M, Saito Y, Suzuki H, Wolff LF, Yoshie H. Platelet-rich plasma contains high levels of platelet-derived growth factor and transforming growth factor-beta and modulates the proliferation of periodontally related cells in vitro. J Periodontol. 2003 Jun;74(6):849-57. doi: 10.1902/jop.2003.74.6.849. PMID 12886996
- [Background] Kawase T, Okuda K, Saito Y, Yoshie H. In vitro evidence that the biological effects of platelet-rich plasma on periodontal ligament cells is not mediated solely by constituent transforming-growth factor-beta or platelet-derived growth factor. J Periodontol. 2005 May;76(5):760-7. doi: 10.1902/jop.2005.76.5.760. PMID 15898937
- [Background] Whitman DH, Berry RL, Green DM. Platelet gel: an autologous alternative to fibrin glue with applications in oral and maxillofacial surgery. J Oral Maxillofac Surg. 1997 Nov;55(11):1294-9. doi: 10.1016/s0278-2391(97)90187-7. PMID 9371122
- [Background] Marx RE. Platelet-rich plasma: evidence to support its use. J Oral Maxillofac Surg. 2004 Apr;62(4):489-96. doi: 10.1016/j.joms.2003.12.003. No abstract available. PMID 15085519
- [Background] Zehnder JL, Leung LL. Development of antibodies to thrombin and factor V with recurrent bleeding in a patient exposed to topical bovine thrombin. Blood. 1990 Nov 15;76(10):2011-6. PMID 2242423
- [Background] Rapaport SI, Zivelin A, Minow RA, Hunter CS, Donnelly K. Clinical significance of antibodies to bovine and human thrombin and factor V after surgical use of bovine thrombin. Am J Clin Pathol. 1992 Jan;97(1):84-91. doi: 10.1093/ajcp/97.1.84. PMID 1728869
- [Background] Mellonig JT. Decalcified freeze-dried bone allograft as an implant material in human periodontal defects. Int J Periodontics Restorative Dent. 1984;4(6):40-55. No abstract available. PMID 6396269
- [Background] Guillemin MR, Mellonig JT, Brunsvold MA. Healing in periodontal defects treated by decalcified freeze-dried bone allografts in combination with ePTFE membranes (I). Clinical and scanning electron microscope analysis. J Clin Periodontol. 1993 Aug;20(7):528-36. doi: 10.1111/j.1600-051x.1993.tb00402.x. PMID 8354729
- [Background] Committee on Research, Science and Therapy of the American Academy of Periodontology.. Tissue banking of bone allografts used in periodontal regeneration. J Periodontol. 2001 Jun;72(6):834-8. doi: 10.1902/jop.2001.72.6.834. PMID 11453248
- [Background] Froum SJ, Wallace SS, Tarnow DP, Cho SC. Effect of platelet-rich plasma on bone growth and osseointegration in human maxillary sinus grafts: three bilateral case reports. Int J Periodontics Restorative Dent. 2002 Feb;22(1):45-53. PMID 11922217
- [Background] Wiltfang J, Kloss FR, Kessler P, Nkenke E, Schultze-Mosgau S, Zimmermann R, Schlegel KA. Effects of platelet-rich plasma on bone healing in combination with autogenous bone and bone substitutes in critical-size defects. An animal experiment. Clin Oral Implants Res. 2004 Apr;15(2):187-93. doi: 10.1111/j.1600-0501.2004.00980.x. PMID 15008930
- [Background] Aghaloo TL, Moy PK, Freymiller EG. Evaluation of platelet-rich plasma in combination with freeze-dried bone in the rabbit cranium. A pilot study. Clin Oral Implants Res. 2005 Apr;16(2):250-7. doi: 10.1111/j.1600-0501.2004.01075.x. PMID 15777336
- [Background] Sanchez AR, Sheridan PJ, Eckert SE, Weaver AL. Regenerative potential of platelet-rich plasma added to xenogenic bone grafts in peri-implant defects: a histomorphometric analysis in dogs. J Periodontol. 2005 Oct;76(10):1637-44. doi: 10.1902/jop.2005.76.10.1637. PMID 16253084
- [Background] Choi BH, Zhu SJ, Kim BY, Huh JY, Lee SH, Jung JH. Effect of platelet-rich plasma (PRP) concentration on the viability and proliferation of alveolar bone cells: an in vitro study. Int J Oral Maxillofac Surg. 2005 Jun;34(4):420-4. doi: 10.1016/j.ijom.2004.10.018. Epub 2005 Jan 27. PMID 16053853